CLINICAL TRIAL: NCT05335655
Title: Use of Intravenous Dexmedetomidine as an Adjuvant to Extend the Duration of Spinal Anesthesia With Hyperbaric Bupivacaine in Orthopedic Surgery in Hospital Central "Dr. Ignacio Morones Prieto": Double Blind Randomized Trial.
Brief Title: IV Dexmedetomidine in the Duration of Spinal Anesthesia With Hyperbaric Bupivacaine: Double Blind Randomized Trial.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Central "Dr. Ignacio Morones Prieto" (Other)
Responsible Party: Principal Investigator, Liliana Serrano Ibarrola, Principal Investigator, Hospital Central "Dr. Ignacio Morones Prieto"
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 24-CEI-001-20160427
Record Dates: First submitted 2022-03-23; First posted 2022-04-19 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Anesthesia; Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Each patient is assigned to one of the two treatment groups (A of B) according to a computer-generated chart of random numbers. Under standard preanesthetic procedures (non-invasive monitoring, premedication), we blindly administer an IV bolus of dexmedetomidine tittered to 0.5mcg per kilogram (real weight), diluted in 10 ml of 0.9% saline solution during 15 minutes before the spinal block. Once the anesthetic effect is confirmed, we begin a maintenance IV infusion for group A, based on dexmedetomidine 100 mcg diluted in 100 ml of 0.9% saline solution tittered at 0.5 mcg per kilogram per hour (real weight). On the other hand, for group B, we administer the same volume (10 ml) of IV 0.9% saline solution for the initial bolus, and for the maintenance infusion we keep equivalent organoleptic characteristics of simple intravenous 0.9% saline solution as well.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): IV bolus of dexmedetomidine, blindly administered and tittered to 0.5mcg per kilogram (real weight), diluted in 10 ml of 0.9% saline solution during 15 minutes before the spinal block. Once the anesthetic effect is confirmed, the maintenance IV infusion, based on dexmedetomidine 100 mcg diluted in 100 ml of 0.9% saline solution tittered at 0.5 mcg per kilogram per hour (real weight), begins.
  Interventions: Drug: Dexmedetomidine injection
- Group B (Placebo Comparator): IV 10 ml initial bolus of 0.9% saline solution during the 15 minutes before the spinal block. Once de anesthetic effect is confirmed, the maintenance infusion of IV 0.9% saline solution (100 ml in equivalent dosage per hour) begins.
  Interventions: Drug: Sodium Chloride 0.9% infusion

INTERVENTIONS:
Drug: Dexmedetomidine injection — IV initial bolus and trans operative dexmedetomidine infusion.
  Other Names: Precedex infusion
  Arms: Group A
Drug: Sodium Chloride 0.9% infusion — IV initial bolus and trans operative infusion of 0.9% saline solution.
  Other Names: Placebo
  Arms: Group B

SUMMARY:
Introduction: Spinal anesthesia produces sensitive and motor block according to the administered local anesthetic. The total duration of surgical anesthesia depends on the dose, intrinsic properties of the anesthetic, and the use of additional drugs. Dexmedetomidine is an alpha-2 adrenergic agonist that has sedative and analgesic effects. The specific action site in the spinal cord receptors and in the locus coeruleus provide as well hypnotic and sympatholytic characteristics. The combination of spinal anesthesia and intravenous dexmedetomidine is a safe option for hemodynamically stable patients undergoing elective surgery. Material and methods: Double blind randomized trial. The objective is to time and compare the total duration of neuraxial blockade with spinal hyperbaric bupivacaine plus intravenous dexmedetomidine, against hyperbaric bupivacaine by itself. 60 patients shall be included, between the ages of 18 and 65 years, classified by the American Society of Anesthesiologists (ASA) I and II, undergoing lower limb elective orthopedic procedure, with spinal anesthesia plus epidural catheter. 50% of the patients (group A) will receive spinal hyperbaric bupivacaine and IV dexmedetomidine at 0.5 mcg/kg (real weight), and the other 50% (group B) will receive spinal hyperbaric bupivacaine plus IV 0.9% saline solution in equivalent volume.

DETAILED DESCRIPTION:
Neuraxial blockade is produced by interrupting nervous impulse transmission with the administration of a local anesthetic. When the drug in injected directly into the subarachnoid space, it passes through the pia mater and enters the Virchow-Robin orifices all the way to the nerve ganglion of the deepest dorsal roots. This nerve endings are highly accessible and easily anesthetized, even with a low dose of local anesthetic, in comparison with the extradural nerves. The speed of the spinal blockade depends on the size, surface, and degree of myelination of the fibers exposed to the anesthetic. However, the regression or termination of the desired effect appears because of the decrease in drug concentration within the cerebrospinal fluid, which happens when the blood vessels inside the pia mater absorb the substances into the systemic circulation to be metabolized and excreted. The rate of elimination depends on the distribution of local anesthetic; while the diffusion surface is larger, the drug exposure to the vessels increases, and thus the time of action will be shorter.

Bupivacaine is one of the most used local anesthetics for spinal anesthesia, with high protein binding and a slow onset because of it relatively elevated pKa. The standard doses for clinical practice make it appropriate for surgical procedures that take 2.5 to 3 hours. The administration of complementary drugs such as dexmedetomidine altogether with the local anesthetic allows a reduction in the dosage, as well as in the requirements for analgesics and sedative drugs along the procedure and through the first hours of the postoperative period.

Dexmedetomidine properly carries its mechanism of action in the pre and post synaptic alpha-2 receptors along the dorsal horn of the spinal cord, decreasing the release of neurotransmitters and thus the pulsatile transmission of impulses. On the other hand, when administered as an IV infusion, this alpha agonist has shown the ability to reach light sedation levels, easily reversed by verbal or tactile stimulus. When acting at the locus coeruleus presynaptic spots, the effect of trans and postoperative analgesia can also be consistently observed. Because of these characteristics, the benefits of intravenous dexmedetomidine have been recently tested over the length and quality of spinal anesthesia with local anesthetics, by being administered as bolus and then as maintenance infusion at variable doses per kilogram.

This therapeutic alternative has been applied during several types of infraumbilical surgeries, such as varicocelectomy, hernioplasty, orchiectomy, and lower limb interventions, without the risk of producing nausea, vomiting, headache, or shivering. The use of this adjuvant provides longer lasting nervous blockade, as well higher time for postoperative analgesia, which helps to reduce the consumption of sedative drugs and opioids since the beginning of the intervention until up to the following first 24 hours. Finally, the undesired effects that have been reported in some populations when receiving this drug (hypotension and bradycardia), appear unfrequently and can be easily reversed with the use of common prescription hemodynamic drugs (atropine, ephedrine).

However, it is common to observe differing therapeutic responses following drug administration during daily clinical practice, which can be often attributed to interindividual differences in drug pharmacokinetics, linked to race, ethnicity, and social habits, that can develop enzymatic variations or genetic polymorphisms. Currently, there are many bibliographic references that support the theories that punctually describe these changes in pharmacological responses between ethnic groups, which is why there is a constant need for testing the efficacy and safety of certain drugs, to improve patient safety and clinical outcomes in all the medical fields.

In this case, the objective of our trial is to evaluate the clinical response to the therapeutic scheme based on intravenous dexmedetomidine added to spinal anesthesia. We expect to determine if this drug could and should be considered regularly as an adjuvant to prolong the duration and improve the anesthetic and analgesic conditions of neuraxial blockade with intrathecal bupivacaine in orthopedic lower limb surgery.

ELIGIBILITY:
Inclusion Criteria:

* Previously accepted and signed informed consent.
* Age between 18 and 65 years
* Male or female
* ASA classified I or II
* Undergoing elective lower limb orthopedic surgery
* Neuraxial anesthesia with 10 mg of spinal bupivacaine (2ml at 0.5%)
* Inert epidural catheter

Exclusion Criteria

* Basal heart rate lower than 55 beats per minute
* Basal mean arterial pressure (MAP) lower than 65 mmHg
* Non-compensated heart disease
* Sinus bradycardia
* Drug allergy or intolerance
* Contraindication for neuraxial blockade

  * Coagulopathy
  * Lumbar structural pathology and/or vertebral instrumentation
  * Local active infection at punction site
  * Thrombocytopenia (lower than 80 K platelets)
  * Non-controlled psychiatric disease
  * Patients that receive drugs such as NSAIDs, acetaminophen and/or opioids within less than 3 hours prior to the procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-06-10 (Estimated); Study Completion 2022-06-15 (Estimated)

PRIMARY OUTCOMES:
Total time of spinal anesthesia with hyperbaric bupivacaine | Up to 300 minutes
  Time (minutes) from anesthetic onset, until first sign (sensitive/motor) of blockade regression.
Presence of post-operative pain | Up to 120 minutes
  Patient refers pain (Yes or No)

SECONDARY OUTCOMES:
Adverse effects Adverse Effects | Through anesthetic period while administering IV drug
  Hypotension and/or Bradycardia during drug infusion

CONTACTS AND LOCATIONS:
Overall Officials: Juan Francisco Hernández Sierra, M in C, Study Director — Universidad Autonoma de San Luis Potosí
Locations (1):
- Hospital Central Dr Ignacio Morones Prieto, San Luis Potosí City, Mexico

IPD SHARING:
Plan to Share IPD: No